CLINICAL TRIAL: NCT02882035
Title: Opioid Free Anesthesia: What About Patient Comfort?
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Université Libre de Bruxelles (Other)
Collaborators: Jules Bordet Institute (Other)
Responsible Party: Principal Investigator, Sarah Saxena, M.D., Université Libre de Bruxelles
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: CE2261
Record Dates: First submitted 2016-08-24; First posted 2016-08-29 (Estimated); Last update posted 2016-08-29 (Estimated); Status verified 2016-08

CONDITIONS: Anesthesia
Keywords: pain; patient comfort
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- OFA (opioid free anesthesia) (Experimental): All drugs were given IV. Induction in the opioid free group began with a loading dose of clonidine (0.2 mcg kg-1), a bolus of ketamine (0.3 mg kg -1) lidocaine (1.5 mg kg -1) and a bolus of propofol (2-3 mg kg -1).
  General anesthesia was maintained with sevoflurane (MAC: 1) (adapted according to hemodynamic stability).
  Upon the incision, acetaminophen (1000 mg) and diclofenac (75 mg) were given in both groups. A bolus of ketamine (0.2mg kg -1) was given if necessary in the opioid free group (up to three bolus max. were permitted).
  A bolus of piritramide (0.03 mg kg -1) was administered upon subcutaneous closure.
  Postoperative pain was treated with IV acetaminophen (1000 mg) every 6 h for the first 24 hours and IV diclofenac (75 mg) every 12 h for the first 24 hours. Patients received a PCIA (patient-controlled intravenous analgesia) pump of piritramide.
  Interventions: Other: OFA
- OA (opioid anesthesia) (No Intervention): All drugs were given IV. Induction in the opioid group began with remifentanil TCI, a bolus of ketamine (0.3 mg kg -1) lidocaine (1.5 mg kg -1) and a bolus of propofol (2-3 mg kg -1).
  General anesthesia was maintained with sevoflurane (MAC: 1). Upon the incision, acetaminophen (1000 mg) and diclofenac (75 mg) were given in both groups.
  A bolus of piritramide (0.03 mg kg -1) was administered upon subcutaneous closure.
  Postoperative pain was treated with IV acetaminophen (1000 mg) every 6 h for the first 24 hours and IV diclofenac (75 mg) every 12 h for the first 24 hours. Patients received a PCIA (patient-controlled intravenous analgesia) pump of piritramide.

INTERVENTIONS:
Other: OFA
  Arms: OFA (opioid free anesthesia)

SUMMARY:
66 female patients undergoing breast cancer surgery were randomized in the Jules Bordet Institute, the Belgian oncology institute. One group received an opioid anesthesia, the other group an opioid free one. The hypothesis of this study was that opioid free anesthesia improves the postoperative quality of recovery of anesthesia.

DETAILED DESCRIPTION:
Opioids used as part of balanced anesthesia have known undesired side effects such as: respiratory depression, post-operative nausea and vomiting, pruritus, difficulty voiding and ileus.

The purpose of this study was to determine whether opioid free anesthesia influences the quality of recovery. A multimodal approach combining ketamine, lidocaine and clonidine was used as an alternative for an opioid based anesthesia.

The hypothesis of this study was that patient comfort and satisfaction level after an opioid free anesthesia would be higher compared to after a more traditional opioid anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Oncological patients undergoing a total mastectomy or lumpectomy associated with a total axillary dissection were screened.
* Patients with an ASA physical status of II were included.
* Knowledge of either French, English or Dutch was required.

Exclusion criteria were the following:

* Allergy or contraindications to one of the study drugs, renal failure, hepatic failure, hyperthyroidism, AV block 2 or 3 or severe bradycardia, left ventricular failure, unstable blood pressure, epilepsy and psychiatric disturbance.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2014-09; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
QoR-40 | 24 hours post-operatively
  Patient comfort was assessed via the QoR-40 questionnaire 24hours post-operatively.

SECONDARY OUTCOMES:
Post-operative NRS | during 24 hours post-operative
  Pain assessment via NRS
Post-operative piritramide consumption | during the first 24 hours post-operative

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Jules Bordet, Brussels, Brussels Capital, Belgium

IPD SHARING:
Plan to Share IPD: Undecided